CLINICAL TRIAL: NCT05693766
Title: Integrating Gene Signatures to Guide HR+MBC Therapy in a Diverse Cohort (INSIGHT)
Brief Title: Gene Signatures to Guide HR+MBC Therapy in a Diverse Cohort
Acronym: INSIGHT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sonya Reid (Other)
Collaborators: Agendia (Industry); Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor-Investigator, Sonya Reid, Assistant Professor of Medicine, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICCBRE2256
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Invasive Mammary Carcinoma; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physician's Choice of Endocrine-based Therapy_Non-Luminal A subtypes (Active Comparator)
  Interventions: Other: Endocrine-therapy; Other: MammoPrint ® and BluePrint assays
- Capecitabine_Non-Luminal A subtypes (Experimental)
  Interventions: Drug: Capecitabine; Other: MammoPrint ® and BluePrint assays

INTERVENTIONS:
Drug: Capecitabine — 2000 mg taken by mouth twice daily for 7 days on, 7 days off
  Arms: Capecitabine_Non-Luminal A subtypes
Other: Endocrine-therapy — Endocrine therapy administered
  Arms: Physician's Choice of Endocrine-based Therapy_Non-Luminal A subtypes
Other: MammoPrint ® and BluePrint assays — Archival tissue will be analyzed using the MammoPrint ® and BluePrint assays

SUMMARY:
This is an open-label, multicenter, two-arm Phase II clinical trial that will evaluate the impact of 2nd line chemotherapy (i.e. capecitabine) on survival in patients with non-Luminal A hormone receptor-positive (HR+) metastatic breast cancer (MBC)

DETAILED DESCRIPTION:
Primary Objective:

- Determine the impact of early chemotherapy (i.e., capecitabine) versus endocrine therapy-based regimen on anti-tumor effect in patients with non-Luminal A hormone receptor-positive (HR+) metastatic breast cancer

Secondary Objectives:

* Compare the safety and tolerability of capecitabine versus endocrine therapy in patients with non-Luminal A hormone receptor-positive (HR+) metastatic breast cancer
* Determine the impact of early chemotherapy (i.e., capecitabine) versus endocrine therapy-based regimen on anti-tumor effect in patients with non-Luminal A hormone receptor-positive (HR+) metastatic breast cancer

Correlatives:

* Determine if the tumor mutations detected in cfDNA are early surrogates of response
* Determine if the cfDNA results at disease progression show new genomic alterations potentially associated with resistance to therapy

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent.
* Subjects ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Clinical stage IV invasive mammary carcinoma or unresectable locoregional recurrence of invasive mammary carcinoma that is:

  * ER (>/=1%) and/or PR (>/= 1%) by IHC and HER2 negative (by IHC or FISH)
* Previously exposed to an aromatase inhibitor (AI) or a selective estrogenreceptor modulator/ downregulator (SERM; SERD) + a CDK4/6 inhibitor.
* Prior radiation permitted (if completed at least 2 weeks prior to study entry. Patients who have received prior radiotherapy must have recovered from toxicity (≤ grade 1) induced by this treatment (except for alopecia)
* Patients with brain metastasis secondary to breast cancer and clinically stable for more than 4 weeks from completion of radiation treatment and off steroids
* Evaluable disease (measurable or non-measurable)

  * Measurable disease, ie, at least 1 measurable lesion as per RECIST 1.1 (a lesion at a previously irradiated site may only be counted as a target lesion if there is clear sign of progression since the irradiation)
  * Patients with bone only disease allowed if possible to evaluate on radiological exams (eg.bone scan, PET/CT, CT, MRI) even if lesions are non-measurable according to RECIST1.1.
* Adequate organ function including:

  * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
  * Platelets ≥ 100 × 10^9/L
  * Hemoglobin ≥ 8/g/dL (may have been transfused)
  * Total serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
  * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 2.5 × ULN (or ≤ 5 × ULN if liver metastases are present)
  * Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 50mL/min as calculated using the Cockcroft-Gault (CG) equation
* For randomized patients only: tumors must be diagnosed as non-Luminal A using the Blueprint® and Mammaprint® tests

Exclusion Criteria:

* Prior chemotherapy in the metastatic setting
* Previous malignant disease other than breast cancer within the last 2 years with associated competing risk, with the exception of basal or squamous cell carcinoma of the skin, cervical carcinoma in situ, or low-risk cancers considered curatively treated (i.e. complete remission achieved at least 2 years prior to first dose of study drugs AND additional therapy not required while receiving study treatment).
* Persisting symptoms related to prior therapy that has not reduced to Grade 1 [National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 5.0]; however, menopausal symptoms, alopecia, and sensory neuropathy Grade ≤ 2 is acceptable
* Pregnant or breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2037-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Up to 3 years

SECONDARY OUTCOMES:
Overall survival at 2 years | Up to 2 years
Overall survival at 5 years | Up to 5 years
Overall survival at 10 years | Up to 10 years
Clinical Benefit Rate | Approximately 6 months
  Percentage of patients without disease progression at 6 months
Overall response rate | Up to 3 years
Incidence of adverse events | Up to 28 days post-treatment
Overall impact of treatment toxicity | Up to 3 years
  Will be measured using Functional Assessment of Cancer Therapy (FACT)-G (5 point Likert-type scale from 1 ("none at all") to 5 ("very much")

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Reid, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (3):
- United States (3):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas

DOCUMENTS (1):
  • Informed Consent Form (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT05693766/ICF_000.pdf